CLINICAL TRIAL: NCT01490307
Title: A Family Intervention for Adolescent Problem Behavior
Brief Title: A Family Intervention for Adolescent Problem Behavior (AKA Project Alliance 2)
Acronym: PAL-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA018374 (NIH); R01DA018374 (NIH)
Record Dates: First submitted 2011-08-16; First posted 2011-12-12 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Substance Use; Conduct Disorder; Depression; Anxiety
Keywords: parenting intervention; Family Check-Up; Anxiety Disorders; Depression; Depressive Disorder; Conduct Disorder; Mental Disorders; Behavioral Symptoms; Mood Disorders; Mental Disorders Diagnosed in Childhood; Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders; Conduct Disorder; Depression; Anxiety Disorders; Depressive Disorder; Mental Disorders; Behavioral Symptoms; Mood Disorders; Neurodevelopmental Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FCU offered (Experimental)
  Interventions: Behavioral: Family Check-Up
- No feedback or services offered (No Intervention)

INTERVENTIONS:
Behavioral: Family Check-Up — The Family Check-Up starts with a rapport-building session that allows therapists to gauge parents' concerns and motivation for change. This is followed by a thorough assessment of individual family strengths and weaknesses, utilizing parent and child questionnaires and family video observations. Parents then receive feedback on the results of the assessment using motivational interviewing techniques. Attention is focused on parents' and children's readiness to change, as well as the delineation of specific change options. Families may continued to receive tailored intervention services using the Everyday Parenting Curriculum.
  Other Names: Adolescent Transitions Project (ATP); Ecological Family Intervention and Treatment (EcoFIT)
  Arms: FCU offered

SUMMARY:
The goal of this project is to empirically refine and improve a comprehensive family-centered prevention strategy for reducing and preventing adolescent substance use and other problem behaviors. This project builds on 15 years of programmatic research underlying the development of the Family Check-up model (FCU), originally referred to as the Adolescent Transitions Program (ATP; Dishion & Kavanagh, 2003), but later expanded as a general approach to mental health treatment for children from ages 2 through 17 (Dishion & Stormshak, 2007). The FCU model is a multilevel, family-centered strategy delivered within the context of a public school setting that comprehensively links universal, selected, and indicated family interventions. Previous research and the investigators' practical experience working in school settings indicate that the intervention strategy needs improvement in 3 critical areas to build on previous significant effects and to enhance the potential for future dissemination and large-scale implementation:(a) improve the feasibility of both the universal level and the indicated level of the intervention by broadening the intervention components and systematically embedding these components into the current behavioral support systems in the schools; (b) address the transition from middle school to high school, with special attention to academic engagement and reduction of deviant peer clustering; and (c) explicitly incorporate principals of successful interventions with families and young adolescents of diverse ethnic groups into both the universal and indicated models. An additional general goal of this study is to develop, test, and refine a set of research-based instruments that facilitate evaluation, training, implementation, and monitoring of intervention fidelity to maximize the potential success of implementation and large-scale dissemination.

Participants include 593 youth and their families recruited from the 6th grade in three public middle schools in Portland, OR. Families were randomly assigned to receive either the FCU intervention model or treatment as usual. Assessments were collected for 5 years through the 10th grade. High school transition planning and intensive intervention efforts occurred in Grades 7-9.

The investigators tested the hypothesis that the FCU intervention will reduce the growth of problem behavior and substance use through the enhancement of family management and parent involvement in school.

DETAILED DESCRIPTION:
Specific aims of the current project are to:

1. Establish a Family Resource Center (FRC) that builds on school-wide behavior management;
2. Extend the intervention model to explicitly address the high school transition;
3. Develop intervention components specifically focused on the cultural enhancement with a broader youth population, and test the efficacy of these interventions for reducing risk and enhancing positive adjustment for youth and their families;
4. Evaluate the preventive impact of family engagement on individual differences in the growth of deviant peer involvement, antisocial behavior, and tobacco, alcohol, and marijuana use during the critical transition to high school; and
5. Develop a training and fidelity model related to change.

ELIGIBILITY:
Inclusion Criteria:

Parents of all sixth grade students across 2 cohorts at 3 public middle schools were invited to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 593 (Actual)
Dates: Start 2006-02; Primary Completion 2010-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
growth in substance use | 5 time points (6th grade, 7th grade, 8th grade, 9th grade, and 10th grade). Avg time between t1 and t2 was 15.1 mo.; avg time between t2 and t3 was 11.9 mo.; avg time between t3 and t4 was 11.4 mo.; avg time between t4 and t5 was 11.6 mo.
  The Student Survey was collected from all youth, regardless of treatment condition, annually across 6th-10th grades. It includes 6 questions about the frequency with which the adolescent used 5 substances in the last month: cigarettes, chewing tobacco or snuff, alcohol (overall quantity and most at one time), marijuana or hashish, and other hard drugs. Growth curve modeling will be used to represent change in substance use across time.
growth in antisocial behavior | 5 time points (6th grade, 7th grade, 8th grade, 9th grade, and 10th grade). Avg time between t1 and t2 was 15.1 mo.; avg time between t2 and t3 was 11.9 mo.; avg time between t3 and t4 was 11.4 mo.; avg time between t4 and t5 was 11.6 mo.
  The Student Survey was collected from all youth, regardless of treatment condition, annually across 6th-10th grades. It includes youth reports of engagement in antisocial behavior during the past month, measured by averaging across 11 items on a 6-point scale ranging from "never" to "more than 20 times" during the past month. The items included content such as lying to parents, staying out all night without permission, stealing, carrying a weapon, and physical aggression. Growth curve modeling will be used to represent change in antisocial behavior across time.
growth in deviant peer involvement | 5 time points (6th grade, 7th grade, 8th grade, 9th grade, and 10th grade). Avg time between t1 and t2 was 15.1 mo.; avg time between t2 and t3 was 11.9 mo.; avg time between t3 and t4 was 11.4 mo.; avg time between t4 and t5 was 11.6 mo.
  The Student Survey was collected from all youth, regardless of treatment condition, annually across 6th-10th grades. It includes youth reports of the behavior of the friends with whom they have spent the most time in the past month. Youth are asked how many of these friends have engaged in 11 behaviors in the past month, using a 5-point scale ranging from "none" to "4 or more." The items include content such as selling illegal drugs, carrying a knife or handgun, and getting arrested. Growth curve modeling will be used to represent change in deviant peer involvement across time.

SECONDARY OUTCOMES:
growth in family management skills | 3 time points (7th grade, summer after 8th grade, and 10th grade). Average time between t1 and t2 was 15.4 months; average time between t2 and t3 was 17.0 months.
  The family assessment was collected from families who received the FCU; it includes caregiver and child assessment packets and parent-child videotaped interactions. Caregiver and child assessments include reports of family management, including parental monitoring and parent-school involvement. Videotaped interactions are evaluated and each family rated on factors such as supervision, listening skills, use of encouragement, and problem solving. Growth curve modeling will be used to represent change in family management skills across time.
positive change in family relationship quality | 3 time points (7th grade, summer after 8th grade, and 10th grade). Average time between t1 and t2 was 15.4 months; average time between t2 and t3 was 17.0 months.
  The family assessment was collected from families who received the FCU; it includes caregiver and child assessment packets and parent-child videotaped interactions. Caregiver and child assessments include reports of positive relationship and family conflict. Videotaped interactions include seven 5-8 minute discussions on family-related matters. These interactions are evaluated and each family rated on positive relationship and family conflict. Growth curve modeling will be used to represent change in family relationship quality across time.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Stormshak, PhD, Principal Investigator — University of Oregon; Thomas J Dishion, PhD, Principal Investigator — University of Oregon; Kathryn A Kavanagh, PhD, Principal Investigator — University of Oregon; Allison S Caruthers, PhD, Study Director — University of Oregon
Locations (1):
- University of Oregon-Child and Family Center, Portland, Oregon, United States

REFERENCES:
- [Derived] Seidman S, Danzo S, Connell A, Stormshak E. The Family Check-Up and Youth Suicide: Assessing Indirect Effects of Improving Self-Regulation and Reducing Depression in Promoting Long-Term Resilience. Suicide Life Threat Behav. 2025 Jun;55(3):e70029. doi: 10.1111/sltb.70029. PMID 40470833